CLINICAL TRIAL: NCT04273464
Title: Secondary Breast Reconstruction in Irradiated Patients - Prospective Trial Comparing DIEP to Brava Expansion + Fat Transplantation
Brief Title: Breast Reconstruction With Autologous Tissue: Microsurgery or Fat Grafting?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1097.13
Record Dates: First submitted 2018-10-29; First posted 2020-02-18 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Mammaplasty
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective comparative study of two parallell cohorts (BRAVA and DIEP reconstruction methods).
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brava-group (Experimental): External tissue expanders will be used 3 weeks prior to operation and 2 weeks postoperatively in order to enhance the volume and survival of fat cells. We expect that each patient in the fat transplantation group will need 4-6 transplantation sessions of about 1.5 to 2 hours each to achieve satisfactory volume and shape of the breast.31 participants.
  Interventions: Procedure: Brava-group
- DIEP-group (Active Comparator): 26 participants. We expect 1-2 operative sessions of respectively 5-7 and 2-3 hours duration in the DIEP group. The risk of reoperation (second operation during the first postoperative week) in the DIEP group is 5-10 %
  Interventions: Procedure: DIEP-group

INTERVENTIONS:
Procedure: Brava-group — Breast reconstruction by external tissue expansion and multiple fat transplantations(Brava group); Breast reconstruction with microsurgical DIEP-flap transfer.
  Arms: Brava-group
Procedure: DIEP-group — Microsurgical reconstruction by DIEPO method
  Arms: DIEP-group

SUMMARY:
Methods for breast reconstruction after mastectomy vary from rather simple techniques using expanders and implants, local flaps alone or in combination with implants, to more complex methods using autologous tissue.Transverse rectus abdominis muscle (TRAM) flap has since 1983 become golden standard in autologous breast reconstruction. The deep inferior epigastric perforator (DIEP)-flap, the very last improvement of TRAM flap, has been used in breast reconstruction after mastectomy and radiation therapy as the method of choice at the Department for Plastic Surgery at Hospital of Telemark since 2000.Transplantation of fat tissue by lipoinjections is an alternative method for partial breast reconstruction. In recent years, fat transplantation techniques have gained interest even for patients after mastectomy, as donor site morbidity and operative trauma seem to be less than when free flaps are used. Best results are obtained if the skin around mastectomy scar is pretreated with external expansion. The results of breast reconstruction with fat transplantation are promising, but have not been compared to microsurgical reconstruction of the breast in a scientific manner. The present project is designed to address clinical questions regarding efficiency and patient satisfaction of the two methods.

DETAILED DESCRIPTION:
When used for breast reconstruction on irradiated patients, breast implants can result in 50% or higher rate of complications included capsular contracture and implant rupture. For this reasons secondary breast reconstruction in irradiated patients is preferably done with autologous tissue.Reconstruction methods employing microvascular transfer of autologous tissue are time consuming having a long learning curve for surgeons. The present project aims to evaluate fat transplantation in combination with external tissue expansion (Brava method) as an alternative to microsurgical complexe methods.

Hypothesis: Early complication/ drop out occur more frequently in fat transplantated patients.

Methods: External tissue expanders (Brava, Brava, LLC 14221 SW 142nd St, Miami, FL 33186) will be used 3 weeks prior to reconstruction in order to enhance the volume and survival of fat cells. The investigators expect that each patient in the fat transplantation group will need 4-6 transplantation sessions of about 1.5 to 2 hours each to achieve satisfactory volume and shape of the breast. The investigators expect 1-2 operative sessions of respectively 5-7 and 2-3 hours duration in the DIEP group. The risk of reoperation (second operation during the first postoperative week) in the DIEP group is 5-10 %.

Patients in the fat transplantation group experiencing poor compliance or early complications as well as patients with unsatisfactory results will be offered alternative methods of reconstruction such as superior or inferior gluteal perforator flap (SGAP or IGAP), Latissimus dorsi pedicled flap alone or in combination with implant. In some cases even simple implant reconstruction could be offered assuming that the quality of previously irradiated skin has been improved by fat transplants .

Study design: Prospective cohort study

Hypothesis: Reconstruction with BRAVA and fat transplantation is a good alternative to reconstruction with DIEP flap.

Study variables: MRI-based volume estimates, anthropometric measurements, VAS scale (Breast-Q - questionnaire measuring patient-related outcome) and Telemark breast score evaluation through independent investigators

Statistics: Power analysis determine that 25 patients are required in each group in this study considering 80 % power with 95 % significance and 40 % difference with regard to patient satisfaction and early complications.

Follow-up: 6 months after DIEP reconstruction and 3 months after the second session of fat transplantation.

Primary endpoint: assessment of early complications in both study groups

Secondary endpoint: patient satisfaction with shape and symmetry of the breast, Satisfaction with psychosocial, psychological and sexual well-being, satisfaction with process of care, shape of the body and postoperative scars (Breast-Q).

ELIGIBILITY:
Inclusion Criteria:

1. Women who have consented to participate in the study and underwent mastectomy and radiation therapy.
2. Mammography of the remaining breast performed within 3 months before surgery
3. At least 1 year after completion of radiotherapy
4. BMI between 22 and 32 -

Exclusion Criteria:

1. Patients with recurrent or metastatic breast cancer
2. Patients with pacemakers or metal clips after any surgery
3. Patients with heart, kidney or liver failure or other medical conditions such as severe hypertension, COPD, autoimmune disorders, SLE or poorly regulated diabetes
4. Patients with claustrophobia
5. Patients with severe drug abuse
6. Patients with silicone allergy
7. Patients with bleeding disorders
8. Patients who smoke or have smoked in the last two months

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Breast-Q reconstructive module | Change in Breast Q score from preop. status(baseline) to 3 months postop.score for Brava group and 6 months for DIEP group
  Patient-related outcome by Breast-Q questionnaire. The Breast-Q™ was developed and provided by the Memorial Sloan Kettering Cancer Center (New York, USA) and the University of British Columbia (Vancouver, British Columbia, Canada). Translation of the BCT Breast-Q™ module into Norwegian was approved in 2014. The questionnaire contains nine domains: satisfaction with breasts, adverse effects of radiation, psychosocial and physical well-being, and different aspects of satisfaction with care. Breast Q preoperative and Breast QQ Breast Q pre- and postoperative scores were registered
Early complications | Three months after first two fat grafting sessions in Brava reonstruction group
  Complications registered in relation to the surgical sessions

SECONDARY OUTCOMES:
Telemark breast score | 3 months after completion of reconstruction for Brava, and 6 months after completion of reconstruction for DIEP-group
  Using the Telemark braest score for assessment of esthetic result

CONTACTS AND LOCATIONS:
Overall Officials: Hege Kersten, PhD, Study Director — Sykehuset Telemark
Locations (1):
- Telemark Hospital, Skien, Telemark, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Begic A, Tolli J, Hegard W, Stark B. Secondary Breast Reconstruction in Irradiated Patients: Prospective Trial Comparing DIEP to Brava Expansion and Fat Transplantation. Plast Reconstr Surg. 2023 Aug 1;152(2):205e-216e. doi: 10.1097/PRS.0000000000010250. Epub 2023 Feb 1. PMID 36723980